CLINICAL TRIAL: NCT02576652
Title: Bone Histomorphometry of the Proximal Femur in Denosumab-treated Subjects Undergoing Total Hip Replacement
Brief Title: Bone Histomorphometry in Postmenopausal Men and Women With Osteoarthritis Undergoing Total Hip Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20140259
Record Dates: First submitted 2015-05-26; First posted 2015-10-15 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Osteoporosis
Keywords: bone biopsy; tetracycline; demeclocycline; total hip replacement
MeSH Terms: conditions — Osteoporosis | interventions — Tetracycline; Demeclocycline; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Osteoarthritis Participants (Other): Participants previously treated with denosumab and planning to undergo total hip replacement (THR) received one cycle of tetracycline administered at either 250 mg four times a day or 500 mg twice a day for 3 days and one cycle of demeclocycline administered at either 150 mg four times a day or 300 mg twice a day for 3 days, ten days after last dose of tetracycline in cycle 1. THR surgery was performed 5 to 42 days after the last dose of demeclocycline.
  Interventions: Other: Tetracycline; Other: Demeclocycline; Procedure: Total Hip Replacement

INTERVENTIONS:
Other: Tetracycline — Treatment during cycle 1 consists of a total oral dose of 1000 mg of tetracycline daily for a total of 3 days.
Other: Demeclocycline — Treatment during cycle 2 consists of a total oral dose of 600 mg of demeclocycline daily for 3 days.
Procedure: Total Hip Replacement — Participants entering this study were prescheduled to undergo elective THR due to osteoarthritis. Surgery was to be performed according to local standard of care. During THR a fragment of femoral bone was acquired for histomorphometry evaluation.

SUMMARY:
The primary objective of this study is to determine the incidence of modeling-based bone formation in the femoral neck in participants who have received denosumab and are undergoing total hip replacement (THR).

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent/assent prior to initiation of any study-specific activities/procedures
* Ambulatory postmenopausal women and men with osteoporosis
* Scheduled to undergo elective THR due to osteoarthritis of the hip
* Received at least 2 doses of denosumab 60 mg subcutaneously over 18 months
* Last dose of denosumab within 6 months of scheduled THR

Exclusion Criteria:

* Received treatment for osteoporosis other than denosumab in one year prior to THR
* Subjects with current diagnosis of any of the following conditions are excluded

  * Current, uncontrolled hypo- or hyperthyroidism (subjects who have controlled hypo- or hyperthyroidism may be eligible, provided that they have been on a stable therapy for at least 3 months [per subject report])
  * Current, hypo- or hyperparathyroidism
  * Osteomalacia
  * Paget's disease of bone
  * Other bone diseases which affect bone metabolism (eg, osteopetrosis, osteogenesis imperfecta)
  * Severe chronic kidney disease (CKD), defined as CKD stage 4 or greater
* Malignancy within the last 5 years (except cervical carcinoma in situ or basal cell carcinoma)
* Self-reported alcohol or drug abuse within the previous 12 months
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s)
* Other investigational procedures while participating in this study are excluded
* Subject has known sensitivity to any of the products to be administered (eg, tetracycline, demeclocycline) during study
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Helen Hayes Hospital, West Haverstraw, New York
  - Research Site, West Haverstraw, New York

REFERENCES:
- [Derived] Dempster DW, Chines A, Bostrom MP, Nieves JW, Zhou H, Chen L, Pannacciulli N, Wagman RB, Cosman F. Modeling-Based Bone Formation in the Human Femoral Neck in Subjects Treated With Denosumab. J Bone Miner Res. 2020 Jul;35(7):1282-1288. doi: 10.1002/jbmr.4006. Epub 2020 Apr 2. PMID 32163613
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one center in the United States.
Groups:
- Osteoarthritis Participants: Participants previously treated with denosumab and planning to undergo total hip replacement (THR) received one cycle of tetracycline administered at either 250 mg four times a day or 500 mg twice a day for 3 days and one cycle of demeclocycline administered at either 150 mg four times a day or 300 mg twice a day for 3 days, ten days after the last dose of tetracycline in cycle 1. THR surgery was performed 5 to 42 days after the last dose of demeclocycline.
Period: Overall Study
Arm/Group | Osteoarthritis Participants
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Osteoarthritis Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Modeling Based Bone Formation in the Femoral Neck
Description: Femoral neck bone samples were prepared according to standard procedures for bone histology and bone histomorphometry at a central bone histomorphometry facility.
  Modeling based formation units in active bone-forming, tetracycline-labeled surfaces were identified by a smooth cement line.
  The percentage of participants with fluorochrome labeling present in the cancellous or periosteal, or endocortical surfaces of the femoral neck indicative of modeling-based bone formation is reported.
Time Frame: Days 22-58 (at the time of hip replacement surgery)
Population: All enrolled participants who had an evaluable biopsy for fluorochrome labeling.
Measure: Number; unit: percentage of participants
Arm/Group | Osteoarthritis Participants
Number analyzed (Participants) | 4
percentage of participants | 100

2. Secondary Outcome: Modeling Based Formation Units in the Femoral Neck
Description: Femoral neck bone samples were prepared according to standard procedures for bone histology and bone histomorphometry at a central bone histomorphometry facility.
  Modeling based formation units in active bone-forming, tetracycline-labeled surfaces were identified by a smooth cement line. The number of modeling based formation units was evaluated at the cancellous, periosteal, and endocortical regions and is reported in units per mm of bone surface.
Time Frame: Days 22-58 (at the time of hip replacement surgery)
Population: Enrolled participants who had an evaluable biopsy for fluorochrome labeling.
Measure: Mean (Standard Deviation); unit: units/mm
Arm/Group | Osteoarthritis Participants
Number analyzed (Participants) | 4
units/mm
  Cancellous Region | 0.1455 (0.2097)
  Endocortical Region | 0.2223 (0.2306)
  Periosteal Region | 0.1990 (0.1409)

3. Secondary Outcome: Overfilled Remodeling-based Formation Units in the Femoral Neck
Description: Femoral neck bone samples were prepared according to standard procedures for bone histology and bone histomorphometry at a central bone histomorphometry facility.
  Remodeling-based formation units in active bone-forming, tetracycline-labeled surfaces were identified by a scalloped cement line. The number of overfilled remodeling-based formation units was evaluated at the cancellous, periosteal, and endocortical regions and is reported as units per mm of bone surface.
Time Frame: Days 22-58 (at the time of hip replacement surgery)
Population: Enrolled participants who had an evaluable biopsy for fluorochrome labeling.
Measure: Mean (Standard Deviation); unit: units/mm
Arm/Group | Osteoarthritis Participants
Number analyzed (Participants) | 4
units/mm
  Cancellous Region | 0.0038 (0.0062)
  Endocortical Region | 0.0108 (0.0138)
  Periosteal Region | 0.0000 (0.0000)

4. Secondary Outcome: Remodeling-based Formation Units Including Overfilled Units in the Femoral Neck
Description: Femoral neck bone samples were prepared according to standard procedures for bone histology and bone histomorphometry at a central bone histomorphometry facility.
  Remodeling based formation units in active bone-forming, tetracycline-labeled surfaces were identified by a scalloped cement line. The number of remodeling based formation units including overfilled units was evaluated at the cancellous, periosteal, and endocortical regions and is reported in units per mm of bone surface.
Time Frame: Days 22-58 (at the time of hip replacement surgery)
Population: Enrolled participants who had an evaluable biopsy for fluorochrome labeling.
Measure: Mean (Standard Deviation); unit: units/mm
Arm/Group | Osteoarthritis Participants
Number analyzed (Participants) | 4
units/mm
  Cancellous Region | 0.0285 (0.0174)
  Endocortical Region | 0.0323 (0.0318)
  Periosteal Region | 0.0033 (0.0065)

ADVERSE EVENTS:
Time Frame: From the date of first administration of fluorochrome treatment (tetracycline or democlocycline or their derivatives) until the date of THP surgery (up to 58 days).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Total Hip Replacement: Participants previously treated with denosumab and planning to undergo THR received one cycle of tetracycline administered at either 250 mg four times a day or 500 mg twice a day for 3 days and one cycle of demeclocycline administered at either 150 mg four times a day or 300 mg twice a day for 3 days, ten days after the receipt of the last dose of tetracycline in cycle 1. THR surgery was performed 5 to 42 days after the last dose of demeclocycline.
Arm/Group | Total Hip Replacement
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Hip Replacement (N=6)
Arthritis infective (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Hip Replacement (N=6)
Hypersensitivity (Immune system disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-11-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT02576652/SAP_000.pdf
  • Study Protocol (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT02576652/Prot_001.pdf